CLINICAL TRIAL: NCT04836572
Title: An Open-label, Non Significant Risk, Adhesive Wear Validation Study for the On Body Drug Delivery Device Component of the SQIN-01 Furosemide Infusor (Infusor Device)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SQ Innovation, Inc. (Industry)
Collaborators: Community Clinical Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SQI-09-01
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer Study
Keywords: Adhesive; Attachment duarability; Assess possible skin reactions; Erythema; Edema
MeSH Terms: conditions — Erythema; Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wear Period (Other)
  Interventions: Other: 3M 1529 Adhesive Tape

INTERVENTIONS:
Other: 3M 1529 Adhesive Tape — 5-12 hour adhesive wear

SUMMARY:
The purpose of the present study is to test the adequacy, performance and skin reactivity of the adhesive tape to be utilized in the to-be-marketed Device.

The present study will examine adhesive hold performance, re-use protection (i.e. adhesive re-application) and skin reactivity/tolerability of the proposed commercial adhesive tape (i.e. within the Test Infusor Device; TID). As the purpose of the study is to assess adhesive performance which does not require activation of the device. Hence in this study no canula will be deployed (no skin penetration) and no delivery of the drug or other fluids.

DETAILED DESCRIPTION:
An open-label, non significant risk, adhesive wear validation study with 60 adult subjects.

Group A (30 subjects): Wearing of the Infusor for 5-9hrs followed by assessment and subsequent removal of the Infusor by study staff with photographic recording prior to and after removal.

Group B (30 subjects): Wearing of the Infusor for 5-9hrs followed by assessment and photographic recording of the Infusor by study staff after which the subject will return home and removal of the Infusor by subject or caregiver approximately 12hrs after placement (± 1hr), when another photograph will be taken. The subject must return the device to the site and transfer the photograph in accordance with the instructions.

Until enrollment for Group B is complete, study candidates will be asked if prefer group A or B. Additional inclusion criteria apply for participation in group B.

Consent, screening and enrollment may be performed on the same day (Day 1) Screening must be performed within 7 days of the Wear phase.

Following signing of the ICF (A or B) each subject will complete Screening activities (height, weight, brief medical history). If the subject meets all inclusion criteria an none of the exclusion criteria the subject may enroll.

The Wear Phase consists of one (1) wear period of five to twelve (5-12) hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be considered for inclusion only if they meet all of the following criteria:

  1. An Institutional Review Board (IRB)-approved informed consent is signed and dated prior to any study-related activities.
  2. Male and female subjects ≥40 and ≤80 years of age
  3. Body mass index (BMI) <38 kg/m2.
  4. Females will be non-pregnant and non-lactating.
  5. Able to participate in the study in the opinion of the Investigator.
  6. Has the ability to understand the requirements of the study and is willing to comply with all study procedures.

Exclusion Criteria:

* Subjects will be excluded from participation if they meet any of the following criteria:

  1. Systolic blood pressure (SBP) <90 mmHg.
  2. Temperature ≥38°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment.
  3. History of COVID-19 infection or recent exposure to someone with COVID-19 or who is currently in quarantine for COVID-19 exposure.
  4. Presence of signs or symptoms of possible COVID-19 infection, including cough, shortness of breath, or temperature ≥ 38°C.
  5. Previous abdominal surgery resulting in presence of a scar or malformation in upper abdominal area.
  6. Presence of skin disorder or abnormality in upper abdominal area.
  7. Known or suspected allergy to acylate adhesives or other materials present in the device.
  8. Significant comorbidities or health issues which in the opinion of the investigator may interfere with study participation or study assessments.
  9. Major surgery within 30 days prior to Screening.
  10. Administration of an investigational drug or implantation of investigational device, or participation in another interventional trial, within 30 days prior to Screening.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Adhesion | 5-9 hours
  Number of participants with failed adhesion (Adhesion Score of 3 or 4 - Appendix A) 5-9 hours after placement as determined by study staff and documented by photography.
Re-adhesion | > 5 hours
  Number of participants with successful re-adhesion - score of 0, 1 or 2 as per Appendix A at 5 minutes after adhesion at the opposite side of the upper abdomen after a completed simulated wear period of no less than 5 hours

SECONDARY OUTCOMES:
Comfort of Wear | 5-12 hours
  Overall average comfort of wear score of the test device using a 10-point Visual Analogue Scale (VAS). The scores are values 0-10, with 0 being very comfortable, and 10 being intolerable discomfort.
Interference | 5-12 hours
  Overall average scoring of interference with important routine activities of daily living such as use of the bathroom, walking, and climbing stairs using a 10-point Visual Analogue Scale (VAS). The scores are values are 0-10, with 0 being no interference, and 10 being great interference.
Irritation | 5-12 hours
  Overall average irritation score for erythema and edema (on a 5-point scale) after wear(Appendix C). The scores are values 0-4 with 0 being no erythema/edema, and 4 being severe erythema/edema.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Magner, RN, Principal Investigator — Community Clinical Research Network
Locations (1):
- Community Clinical Research Network, Marlborough, Massachusetts, United States